CLINICAL TRIAL: NCT07135596
Title: Research on the Effectiveness and Safety of Treatment With OviTex® PRS - a Breast Reconstruction Evaluation
Brief Title: Effectiveness and Safety of OviTex® PRS in Breast Reconstruction
Acronym: RESTORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tela Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TB_05
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- OviTex PRS (Experimental)
  Interventions: Device: OviTex PRS

INTERVENTIONS:
Device: OviTex PRS — A multi-layer construct of extracellular matrix (ECM) derived from ovine forestomach and embroidered with polymer filament.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of OviTex PRS in subjects undergoing implant-based breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a female between the ages of 22 - 75, inclusive, at the time of enrollment (e.g. date of index surgical procedure);
2. Patient is planned for a first-time immediate unilateral or bilateral DTI pre-pectoral breast reconstruction following mastectomy for cancer or as cancer prophylaxis;
3. Patient is not a current cigarette smoker;
4. Patient is willing and able to voluntarily sign the IRB approved Subject Informed Consent Form;
5. Patient is willing and able to comply with the study requirements including completion of required follow-up visits, subject questionnaires, clinic evaluations, and photographs.

Exclusion Criteria:

1. Patient has a BMI < 18.5 or > 35;
2. Patient is undergoing radical mastectomy;
3. Breast reconstruction plan includes hybrid implant coverage using another type of mesh (synthetic or ADM) or another autologous treatment such as large latissimus flap, abdominal flap or similar;
4. Breast reconstruction plan includes a custom sized breast implant, permanent breast implant greater than 800cc, and/or a permanent breast implant that is not FDA approved for use in breast reconstruction;
5. Patient has undergone prior breast reconstruction, breast augmentation, mastopexy, or breast reduction surgeries (not including breast biopsy);
6. Patient is undergoing delayed reconstruction;
7. Patient has received neo-adjuvant radiation to the chest (including any previous history of whole breast radiation or mantle radiation);
8. Patient has received neo-adjuvant chemotherapy within the 4 weeks prior to enrollment;
9. Patient has received Keytruda therapy or is planning to receive Keytruda therapy during study participation;
10. Patient has uncontrolled Type I or Type II diabetes (HbA1C >7%);
11. Patient is pregnant or planning to become pregnant during study participation and up to 5 years from the index surgical procedure;

    • If the subject is not post-menopausal, agree to take adequate birth control precautions during study participation;
12. Patient has been diagnosed with a medical condition or is taking medications which are known to impact wound healing, weaken the body's natural resistance to disease, result in elevated postoperative risks, or may otherwise affect the validity of the study;
13. Patient has a known sensitivity or allergy to poly(lactic-co-glycolic acid) (PLGA) or materials of ovine (sheep) origin;
14. Patient is diagnosed with a bleeding disorder in which medication is not stopped within 2 weeks of the index procedure;
15. Patient is currently diagnosed with drug or alcohol abuse or has a known history with relapse within the past 3 years;
16. Patient is currently participating in another drug or device clinical trial;
17. Patient is currently imprisoned.

Intraoperative Exclusion Criteria

All subjects will be evaluated intraoperatively for the following exclusion criteria:

1. Subject does not receive an immediate pre-pectoral direct-to-implant breast reconstruction;
2. Study device will not be used during the procedure or a non-eligible device will be implanted.

Ages: 22 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Reconstructive Failure Rate | From enrollment to 12 months
Major Complication Rate | From enrollment to 12 months

IPD SHARING:
Plan to Share IPD: No